CLINICAL TRIAL: NCT00144417
Title: TBTC Study 28: Evaluation of a Moxifloxacin-based, Isoniazid-sparing Regimen for Tuberculosis Treatment
Brief Title: TBTC Study 28: Moxifloxacin Versus Isoniazid for TB Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Global Alliance for TB Drug Development (Other); Bayer (Industry)
Responsible Party: Dr. Stefan Goldberg, CHSRB/DTBE/NCHHSTP/CDC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-4448
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-06

CONDITIONS: Tuberculosis
Keywords: tuberculosis; TB; treatment; efficacy; safety
MeSH Terms: conditions — Tuberculosis | interventions — Moxifloxacin; Pyrazinamide; Ethambutol; Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HRZE (Active Comparator): isoniazid, rifampin, pyrazinamide, ethambutol, moxifloxacin-placebo
  Interventions: Drug: isoniazid
- MRZE (Experimental): moxifloxacin, rifampin, pyrazinamide, ethambutol, isoniazid-placebo
  Interventions: Drug: Moxifloxacin (with rifampin, pyrazinamide, and ethambutol)

INTERVENTIONS:
Drug: Moxifloxacin (with rifampin, pyrazinamide, and ethambutol) — Moxifloxacin 400mg daily, 8 weeks
  Arms: MRZE
Drug: isoniazid — isoniazid, oral, 300 mg, daily, 8 weeks
  Arms: HRZE

SUMMARY:
This double-blind, randomized controlled trial evaluates moxifloxacin versus isoniazid in daily treatment during the first two months of treatment with rifampin, pyrazinamide and ethambutol for sputum smear-positive pulmonary tuberculosis.

DETAILED DESCRIPTION:
The primary objective of this Phase 2 clinical trial is to compare the safety and antimicrobial activity of a moxifloxacin-containing regimen (moxifloxacin, rifampin, pyrazinamide, ethambutol [MRZE]) in which moxifloxacin has been substituted for isoniazid, to the standard control regimen (isoniazid, rifampin, pyrazinamide, ethambutol [HRZE]) in the first two months of treatment of sputum smear-positive pulmonary tuberculosis. The assessment of antimicrobial activity will be sputum culture-conversion. Higher rates of sputum culture conversion after 2 months of treatment with a moxifloxacin-containing regimen would support Phase 3 clinical trials of moxifloxacin in treatment regimens of less than the current 6 month standard regimens.

Rationale - Current treatment of smear positive pulmonary tuberculosis requires a minimum of 6 months, a treatment duration that is challenging for patients and tuberculosis control programs. Therefore, a high priority in tuberculosis research is the identification of agents that can shorten treatment. Several fluoroquinolone antibiotics have potent activity against Mycobacterium tuberculosis (M. tuberculosis) in preclinical testing. Of the currently available fluoroquinolones, moxifloxacin has excellent activity in vitro and in animal models of tuberculosis, a favorable pharmacokinetic profile (serum half-life of 10-12 hours), lack of problematic drug-drug interactions, no need for dosage adjustment for renal and hepatic insufficiency, and an excellent safety profile. In addition, in the murine model of tuberculosis, the substitution of moxifloxacin for isoniazid resulted in significant reductions in the time to culture conversion and the time to sterilization when compared to the standard combination rifampin, isoniazid and pyrazinamide. However, moxifloxacin has not been fully evaluated in humans for tuberculosis treatment. There is a need to assess not only the anti-tuberculosis activity of moxifloxacin-containing regimens, but also the safety of more prolonged therapy with moxifloxacin.

Two-month culture conversion rates are a well-accepted surrogate marker for the sterilizing activity of anti-tuberculosis drugs. Rifampin and pyrazinamide, the key drugs in current 6-month regimens, markedly increase 2-month culture-conversion rates. Therefore, this study will use 2-month culture conversion rate as the measure of antimicrobial activity of moxifloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Suspected pulmonary tuberculosis with acid-fast bacilli in a stained smear of expectorated or induced sputum. Patients whose sputum cultures do not grow M. tuberculosis and those having an M. tuberculosis isolate resistant to (one or more) isoniazid, rifampin, fluoroquinolones, will be discontinued from the study, but followed for 14 days to detect late toxicities from study therapy. Patients having extra-pulmonary manifestations of tuberculosis, in addition to smear-positive pulmonary disease, are eligible for enrollment. Sputum must be expectorated or induced; smear results from respiratory secretions obtained by bronchoalveolar lavage or bronchial wash may not be used for assessment of study eligibility.
* Willingness to have HIV testing performed, if HIV serostatus is not known or if the last documented negative HIV test was more than 6 months prior to enrollment. HIV testing does not need to be repeated if there is written documentation of a positive test (positive ELISA and Western Blot or a plasma HIV-RNA level greater than 5000 copies/ml) at any time in the past.
* 7 (seven) or fewer days of multidrug therapy for tuberculosis disease in the 6 months preceding enrollment.
* 7 (seven) or fewer days of fluoroquinolone therapy in the 3 months preceding enrollment.
* Age > 18 years
* Karnofsky score of at least 60 (requires occasional assistance but is able to care for most of his/her needs; see Appendix B).
* Signed informed consent
* Women with child-bearing potential must agree to practice an adequate (barrier) method of birth control or to abstain from heterosexual intercourse during study therapy.
* Laboratory parameters done at, or <14 days prior to, screening:
* Serum amino aspartate transferase (AST) activity ≤ 3 times the upper limit of normal
* Serum total bilirubin level ≤ 2.5 times the upper limit of normal
* Serum creatinine level ≤ 2 times the upper limit of normal
* Complete blood count with hemoglobin level of at least 7.0 g/dL
* Complete blood count with platelet count of at least 50,000/mm3
* Serum potassium > 3.5 meq/L
* Negative pregnancy test (women of childbearing potential)

Exclusion Criteria:

* Breast-feeding
* Known intolerance to any of the study drugs
* Known allergy to any fluoroquinolone antibiotic
* Concomitant disorders or conditions for which moxifloxacin (MXF), isoniazid (INH), rifampin (RIF), pyrazinamide (PZA), or ethambutol (EMB) are contraindicated. These include severe hepatic damage, acute liver disease of any cause, and acute uncontrolled gouty arthritis.
* Current or planned therapy during the intensive phase of therapy using drugs having unacceptable interactions with rifampin (rifabutin can be substituted for rifampin during the continuation phase of therapy).
* Current or planned antiretroviral therapy during the intensive phase of therapy.
* History of prolonged QT syndrome or current or planned therapy with quinidine, procainamide, amiodarone, sotalol, disopyramide, ziprasidone, or terfenadine during the intensive phase of therapy.
* Pulmonary silicosis
* Central nervous system TB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
• To compare the culture-conversion rate at the end of the intensive phase of therapy of the moxifloxacin regimen vs. that of the isoniazid regimen | 8 weeks

SECONDARY OUTCOMES:
To compare the safety and tolerability of the moxifloxacin regimen to that of the isoniazid regimen | 8 weeks
To determine the time to culture-conversion of the moxifloxacin regimen and the isoniazid regimen using data from 2-, 4-, 6-, and 8-week cultures | 8 weeks
To compare the proportion of patients with any Grade 3 or 4 adverse reactions | 8 weeks
To compare adverse events and 2-month culture conversion rates among HIV-infected patients vs. HIV-uninfected patients | 8 weeks
To compare the rates of treatment failure of the moxifloxacin regimen and the isoniazid regimen | 6 months
To determine whether there is delayed toxicity attributable to moxifloxacin (toxicity that becomes evident after the 8 weeks of moxifloxacin therapy) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Chaisson, MD, Study Chair — Johns Hopkins University; Susan E Dorman, MD, Principal Investigator — Johns Hopkins University; John L Johnson, MD, Principal Investigator — Case Western Reserve University
Locations (26):
- United States (20):
  - Veterans Administration Medical Center of Arkansas, Little Rock, Arkansas
  - University of Southern California Medical Center, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California, San Francincisco, San Francisco, California
  - Denver Public Health Department, Denver, Colorado
  - Washington DC Veterans Administration Medical Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Hines Veterans Administration Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - New Jersey School of Medicine, Newark, New Jersey
  - Columbia University, New York, New York
  - Harlem Hospital, Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Veterans Administration Tennessee Valley Health Care System, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston Veterans Administration Medical Center, Houston, Texas
  - Audie L Murphy Memorial Veterans Administration Medical Center, San Antonio, Texas
  - Seattle-King County Health Department, Seattle, Washington
- Hopital Universitario Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (2):
  - University of Manitoba, Winnepeg, Manitoba
  - Montreal Chest Institute, Montreal, Quebec
- Nelson R. Mandela School of Medicine, Durban, KwaZulu-Natal, South Africa
- Agencia de Salut Publica, Barcelona, Spain
- Makerere University Medical School, Kampala, Uganda

REFERENCES:
- [Result] Dorman SE, Johnson JL, Goldberg S, Muzanye G, Padayatchi N, Bozeman L, Heilig CM, Bernardo J, Choudhri S, Grosset JH, Guy E, Guyadeen P, Leus MC, Maltas G, Menzies D, Nuermberger EL, Villarino M, Vernon A, Chaisson RE; Tuberculosis Trials Consortium. Substitution of moxifloxacin for isoniazid during intensive phase treatment of pulmonary tuberculosis. Am J Respir Crit Care Med. 2009 Aug 1;180(3):273-80. doi: 10.1164/rccm.200901-0078OC. Epub 2009 Apr 30. PMID 19406981
- [Derived] Zhang N, Savic RM, Boeree MJ, Peloquin CA, Weiner M, Heinrich N, Bliven-Sizemore E, Phillips PPJ, Hoelscher M, Whitworth W, Morlock G, Posey J, Stout JE, Mac Kenzie W, Aarnoutse R, Dooley KE; Tuberculosis Trials Consortium (TBTC) and Pan African Consortium for the Evaluation of Antituberculosis Antibiotics (PanACEA) Networks. Optimising pyrazinamide for the treatment of tuberculosis. Eur Respir J. 2021 Jul 20;58(1):2002013. doi: 10.1183/13993003.02013-2020. Print 2021 Jul. PMID 33542052
- [Derived] Mac Kenzie WR, Heilig CM, Bozeman L, Johnson JL, Muzanye G, Dunbar D, Jost KC Jr, Diem L, Metchock B, Eisenach K, Dorman S, Goldberg S. Geographic differences in time to culture conversion in liquid media: Tuberculosis Trials Consortium study 28. Culture conversion is delayed in Africa. PLoS One. 2011 Apr 11;6(4):e18358. doi: 10.1371/journal.pone.0018358. PMID 21494548